CLINICAL TRIAL: NCT06788886
Title: Enhancing Brain and Mental Health Through Respiratory Training: Clinical Applications in Cancer and Neurodegenerative Disease Care for Patients and Caregivers (Breathing Study)
Brief Title: Breathing Practice for Brain and Mental Health in Cancer and Neurodegenerative Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-000979; NCI-2025-00205 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000979 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Malignant Brain Neoplasm; Malignant Solid Neoplasm; Multiple Sclerosis; Neuroendocrine Tumor; Prostate Carcinoma
MeSH Terms: conditions — Brain Neoplasms; Multiple Sclerosis; Neuroendocrine Tumors; Prostatic Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Respiratory Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Study 1 Group 1, Subgroup 1 (6 month breathing sessions) (Experimental): Participants engage in breathing self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Participants then engage in breathing self-practice routines using a mobile app over 30 minutes daily for an additional 2 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Participants also undergo MRI scans throughout the study.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Respiratory Therapy
- Study 1 Group 1, Subgroup 2 (4 month breathing sessions) (Experimental): Participants engage in breathing self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Participants then discontinue breathing self-practice routines for the additional 2 months on study. Participants also undergo MRI scans throughout the study.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Respiratory Therapy
- Study 1 Group 2, Subgroup 3 (6 month walking routines) (Active Comparator): Participants engage in walking self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may also participate in in-person group walking session with other participants weekly on study. Participants then engage in walking self-practice routines using a mobile app over 30 minutes daily for an additional 2 months on study. Participants may also participate in in-person group walking session with other participants weekly on study. Participants also undergo MRI scans throughout the study.
  Interventions: Other: Exercise Intervention; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration
- Study 1 Group 2, Subgroup 4 (walking + breathing) (Experimental): Participants engage in walking self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may also participate in in-person group walking session with other participants weekly on study. Participants then engage in walking self-practice routines using a mobile app over 30 minutes daily for an additional 2 months and also engage in breathing self-practice routines using a mobile app over 30 minutes daily for 2 months on study. Participants may also participate in in-person group walking session with other participants weekly on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Participants also undergo MRI scans throughout the study.
  Interventions: Other: Exercise Intervention; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Respiratory Therapy
- Study 2 (4 month breathing sessions) (Experimental): Cancer patients and their caregivers engage in breathing self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Participants also undergo MRI scans throughout the study.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Respiratory Therapy
- Study 3 Subgroup 5 (6 month breathing sessions) (Experimental): MS patients engage in breathing self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. MS patients then engage in breathing self-practice routines using a mobile app over 30 minutes daily for an additional 2 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Patients also undergo MRI scans and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Respiratory Therapy
- Study 3 Subgroup 6 (4 months breathing sessions) (Experimental): MS patients engage in breathing self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. MS patients then discontinue breathing self-practice routines for the additional 2 months on study. Patients also undergo MRI scans and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Respiratory Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Study 3 Subgroup 5 (6 month breathing sessions); Study 3 Subgroup 6 (4 months breathing sessions)
Other: Exercise Intervention — Participate in walking routines
  Arms: Study 1 Group 2, Subgroup 3 (6 month walking routines); Study 1 Group 2, Subgroup 4 (walking + breathing)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies
Procedure: Respiratory Therapy — Participate in breathing sessions
  Arms: Study 1 Group 1, Subgroup 1 (6 month breathing sessions); Study 1 Group 1, Subgroup 2 (4 month breathing sessions); Study 1 Group 2, Subgroup 4 (walking + breathing); Study 2 (4 month breathing sessions); Study 3 Subgroup 5 (6 month breathing sessions); Study 3 Subgroup 6 (4 months breathing sessions)

SUMMARY:
This clinical trial studies the effect of respiratory training for enhancing brain and mental health among patients with multiple sclerosis (MS) and cancer (along with their caregivers). The relationship between respiration, cardiovascular effects in the brain, mental health, and neurophysiological mechanisms are significant for patient populations facing complex health challenges, such as those with cancer and neurodegenerative disease, and their caregivers. By measuring oxygen delivery to brain tissues and cerebrospinal fluid flow, this trial may help researchers investigate the potential benefits of respiratory training for patients with MS and cancer and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the immediate and long-term effects of improved respiratory function on local tissue oxygen delivery and cerebral circulation, by comparing control and training groups.

SECONDARY OBJECTIVE:

I. To identify key biological aspects of breathing related to brain health and mental well-being, our research explores how respiratory function can improve clinical symptoms related to fatigue and emotional states.

EXPLORATORY OBJECTIVE:

I. To establish a clinically applicable support tool that uses effective breathing practice to help patients, and their caregivers better navigate their clinical treatment.

OUTLINE: Participants are assigned to 1 of 3 studies.

STUDY 1: Participants are randomized to 1 of 2 groups.

GROUP 1: Participants engage in breathing self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. At month 4, participants are randomized to 1 of 2 subgroups.

SUBGROUP 1: Participants engage in breathing self-practice routines using a mobile app over 30 minutes daily for an additional 2 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Participants also undergo MRI scans throughout the study.

SUBGROUP 2: Participants discontinue breathing self-practice routines for the additional 2 months on study. Participants also undergo MRI scans throughout the study.

GROUP 2: Participants engage in walking self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may also participate in in-person group walking session with other participants weekly on study. At month 4, participants are randomized to 1 of 2 subgroups.

SUBGROUP 3: Participants engage in walking self-practice routines using a mobile app over 30 minutes daily for an additional 2 months on study. Participants may also participate in in-person group walking session with other participants weekly on study. Participants also undergo MRI scans throughout the study.

SUBGROUP 4: Participants engage in walking self-practice routines using a mobile app over 30 minutes daily for an additional 2 months and also engage in breathing self-practice routines using a mobile app over 30 minutes daily for 2 months on study. Participants may also participate in in-person group walking session with other participants weekly on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Participants also undergo MRI scans throughout the study.

STUDY 2: Cancer patients and their caregivers engage in breathing self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Participants also undergo MRI scans throughout the study.

STUDY 3: MS patients engage in breathing self-practice routines using a mobile app over 30 minutes daily for 4 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. At month 4, participants are randomized to 1 of 2 subgroups.

SUBGROUP 5: MS patients engage in breathing self-practice routines using a mobile app over 30 minutes daily for an additional 2 months on study. Participants may participate in real-time online breathing sessions with instructors weekly on study. Participants may also participate in in-person breathing sessions with instructors monthly on study. Patients also undergo MRI scans and blood sample collection throughout the study.

SUBGROUP 6: MS patients discontinue breathing self-practice routines for the additional 2 months on study. Patients also undergo MRI scans and blood sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* STUDY 1: Participants must be physically fit enough to perform light exercise.
* STUDY 1: Should read and understand English well enough to consent, complete measures, and follow instructions.
* STUDY 1: Must have access to a smartphone or tablet.
* STUDY 2: Participants must be physically fit enough to perform light exercise.
* STUDY 2: Cancer patients may have prostate cancer, neuroendocrine tumor, or brain cancer in any stage.
* STUDY 2: The main focus is on pairs of cancer patients and their respective caregivers, but individual cancer patients or individual caregivers are also acceptable.
* STUDY 2: Participants should read and understand English well enough to consent, complete measures, and follow instructions.
* STUDY 2: They also must have access to a smartphone or tablet.
* STUDY 3: Participants must be physically fit enough to perform light exercise.
* STUDY 3: The patient should have multiple sclerosis.
* STUDY 3: Participants should read and understand English well enough to consent, complete measures, and follow instructions.
* STUDY 3: They also must have access to a smartphone or tablet.

Exclusion Criteria:

* STUDY 1: Participants incompatible with MRI machines due to factors such as pacemakers or metallic implants.
* STUDY 1: Additionally, those with chronic medical conditions, including heart disease (coronary artery disease, congestive heart failure, hypertension, cardiac arrhythmia), chronic obstructive pulmonary disease (COPD), cystic fibrosis, cancer, diabetes, sleep apnea, aneurysms, and neurological conditions (epilepsy, Alzheimer's disease, Huntington' disease, essential tremor and Parkinson disease) are excluded.
* STUDY 1: Participants with psychiatric conditions such as psychosis, suicidality, bipolar disorder, major depression, and substance use disorders are excluded.
* STUDY 1: Participants serving as caregivers for any of the aforementioned conditions and for other illnesses such as cancer or neurological disorders, are also excluded.
* STUDY 1: Further exclusions apply to those with severe vision, hearing impairments, have a body mass index (BMI) over 30, and those who are pregnant.
* STUDY 1: Those planning to become pregnant during the study period will be excluded.
* STUDY 2: Participants incompatible with MRI machines due to factors such as pacemakers or metallic implants are excluded, as are those with chronic lung disease (chronic obstructive pulmonary disease [COPD], cystic fibrosis), aneurysms, and those who are pregnant.
* STUDY 2: Those planning to become pregnant during the study period will be excluded.
* STUDY 3: Participants incompatible with MRI machines due to factors such as pacemakers or metallic implants are excluded, as are those with chronic lung disease (chronic obstructive pulmonary disease [COPD], cystic fibrosis), aneurysms, and those who are pregnant.
* STUDY 3: Those planning to become pregnant during the study period will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-01-18 (Estimated); Study Completion 2027-01-18 (Estimated)

PRIMARY OUTCOMES:
Changes in respiratory function correlated with brain activity | Baseline up to 6 months
  Assessed using advanced imaging techniques (such as MRI) and physiological analyses. The approach to data analysis will involve a detailed examination of the MRI data collected from each participant. Respiratory data will be correlated with neuroimaging findings to provide a comprehensive view of how respiratory patterns may influence brain activity.

SECONDARY OUTCOMES:
Change in QOL - PHQ-9 | Baseline up to 6 months
  Assessed using the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 consists of 9 questions related to problems experienced over the past 2 weeks. Questions are answered on a scale of 0-3 where 0=Not at all; 1=several days; 2=more than half the days, and 3=nearly every day.
Change in QOL - GAD-7 | Baseline up to 6 months
  Assessed using the Generalized Anxiety Disorder-7 (GAD-7). The GAD-7 consists of 7 questions related to problems experienced over the past 2 weeks. Questions are answered on a scale of 0-3 where 0=Not at all; 1=several days; 2=more than half the days, and 3=nearly every day.
Change in QOL - Linear Analog Self Assessment | Baseline up to 6 months
  Assessed using the Linear Analog Self Assessment, which consists of 5 questions related to feeling related to well being experienced over the past week. Questions are answered on a scale ranging from 0-10 where 0=as bad as it can be and 10=as good as it can be.
Adherence to the breathing protocol for the intention group | Up to 6 months
Change in sleep quality - PSQI | Baseline up to 6 months
  Assessed using the Pittsburgh Sleep Quality Index (PSQI), which consists of questions related to sleep habits during the past month. Questions begin with sleep habits (general time going to bed, how long to fall asleep, general rising time, etc.). These are followed by a list of items answered on scale of 0-3 where 0=not during the past month; 1=less than once a week; 2=once or twice a week ;and 3=three or more times a week. Higher scores indicate worse sleep quality.
Change in sleepiness - ESS | Baseline up to 6 months
  Assessed using the Epworth Sleepiness Scale (ESSI), which consists of questions related to sleep habits during the past month. The survey consists of a list of eight situations in which the respondents rate their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. The scale estimates whether participants are experiencing excessive sleepiness, which higher scores indicating a higher level of sleepiness..
Change in fatigue - MFIS | Baseline up to 6 months
  Assessed using the Modified Fatigue Impact Scale (MFIS), which consists of 21 questions related to the effects of fatigue over the past 4 weeks. Questions are answered on a scale of 0-4 where 0=never; 1=rarely; 2=sometimes; 3=often; and 4=almost always.
Change in caregiver strain - CSI | Baseline up to 6 months
  Assessed using the Caregiver Strain Index (CSI), a list of 13 "things that other people have found to be difficult." Caregivers respond with yes or no to indicate whether each item applies to them.
Change in resilience - BRS | Baseline up to 6 months
  Assessed using the Brief Resilience Scale (BRS), which consists of 6 items answered on a scale of 1-5 where 1=strongly disagree; 2=disagree; 3=neutral; 4=agree, and 5=strongly agree (or the reverse, i.e. 5=strongly disagree and 1=strongly agree). Higher scores generally indicate stronger resilience.
Change in ability to implement health-promoting behaviors - SRAHP | Baseline up to 6 months
  Assessed using the Self Rated Abilities for Health Practices Scale (SRAHP), a 28-item, 5-point scale. SRAHP contains four subscales: Exercise, Nutrition, Responsible Health Practice, and Psychological Well Being. Each subscale has seven items. Respondents are asked to rate the extent to which they are able to perform health practices related to these four domains. Responses are on a 5-point scale where 0=not at all; 1=a little; 2=somewhat; 3=mostly; and 4=completely. Higher scores indicate greater self-efficacy for health practices.

CONTACTS AND LOCATIONS:
Overall Officials: Paul H. Min, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials